CLINICAL TRIAL: NCT06959953
Title: Low-cost Model Versus Airway Part-task Trainer for Flexible Bronchoscope-guided Tracheal Intubation Training: A Multicenter, Non-inferiority, Simulation-based Trial Among Anesthesiology Residents in Lebanon
Brief Title: Low-Cost Model Versus Airway Part-Task Trainer for Flexible Bronchoscope-Guided Tracheal Intubation Training
Acronym: RAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Rony Al Nawar, Doctor in Anesthesiology, Lebanese American University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LebaneseAU
Record Dates: First submitted 2024-11-03; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Simulation Based Medical Education; Tracheal Intubation; Medical Residents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor and the data analyst will be blinded for the allocation arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-cost model (Experimental) (Experimental): In this arm, the residents will train using the locally designed low-cost model that was developed by the study investigator at his institution.
  Here is a short description of the developed model: RAN is a low-cost, locally designed model developed at the investigator's institution using readily available and recyclable materials. This model provides a simulation environment for anesthesiology residents to practice and refine their skills. The primary structure of the training model is fashioned from an old portable 3-drawer organizer unit, repurposed to serve as the foundation for the training apparatus. Utilizing recyclable anesthesia items, including endotracheal tubes (both single lumen and double lumen) with their cuffs, connectors, laryngeal mask airways, oropharyngeal and nasopharyngeal airways, the model replicates the anatomy and equipment encountered during tracheal intubation procedures.
  Interventions: Other: Low-cost model
- Airway part-task trainer (Comparator) (Active Comparator): In this group, the participants will undergo hands-on training using the commercial airway part-task trainer. The commercial airway part-task trainer is the routinely used simulator at the investigator's institution and other institutions as well.
  Interventions: Other: Airway Part-task Trainer

INTERVENTIONS:
Other: Low-cost model — The primary structure of a low-cost training model fashioned from an old portable 3-drawer organizer unit repurposed to serve as the foundation for the training apparatus. This training apparatus will act as the experimental arm to compare it to the Airway Part-Task Trainer in FBTI.
  Other Names: RAN LCM
  Arms: Low-cost model (Experimental)
Other: Airway Part-task Trainer — Training using Airway Part-Task Trainer
  Arms: Airway part-task trainer (Comparator)

SUMMARY:
Background: Awake flexible bronchoscope-guided tracheal intubation (FBTI) is crucial in managing challenging airway situations. As the gold standard for difficult airway management, FBTI is essential for anesthesiologists to navigate anatomical complexities effectively.

Training in FBTI requires theoretical understanding, hands-on practice, and experience. Skill acquisition and knowledge must reach an appropriate level before trainees perform on patients. Simulated scenarios offer a controlled environment for practitioners to develop muscle memory and problem-solving skills without risking patient safety. However, commercial simulators for FBTI are often expensive and inaccessible in many countries. Lebanon, a low- and middle-income country, currently faces a multifaceted economic and financial crisis. Hence, securing enough internal funds to support novice learners using available high-cost simulator training is challenging. Various low-cost simulators have been proposed in the literature, aiming to provide affordable training for novice anesthesiologists, particularly in regions where expensive simulators are scarce.

Aim: This study aims to evaluate a low-cost, locally designed simulator by comparing skill acquisition and retention to a commercial airway part-task trainer in FBTI.

Study design: Multicenter simulation-based randomized controlled trial (RCT) Methods: This simulation-based interventional clinical trial will include anesthesia PGY-I and PGY-II residents inexperienced in FBTI techniques from eight medical schools in Lebanon. The study comprises two main phases and one intermediate phase. Phase one is the development phase, whereby a Delphi approach will be utilized to develop a standardized Global Rating Scale for FBTI (LAU-modified SGR). The intermediate phase constitutes piloting the tool developed with LAU postgraduate trainees years 3, 4, and 5 from the pulmonology department, Ear, Nose, and Throat department, along with the anesthesiology residents. Phase two is the main RCT study whereby all participating residents will receive training on a theoretical course covering flexible bronchoscopy equipment, anatomy, indications, and complications, which will also be supplemented by a procedural video. After which residents will be randomly assigned to one of two groups. One group will undergo training on the locally designed low-cost model (RAN), whereas the other group will train on the airway part-task trainer. Participants' FBTI skills will be assessed using the high-fidelity CAS simulator and the LAU-modified SGR for FBTI to evaluate both theoretical and procedural fluency (i.e., retention of FBTI skills). Assessments will be conducted immediately after the training sessions, with follow-ups at three and six months.

Significance: The utilization of low-cost simulators enables the integration of simulation training for healthcare professionals across diverse settings, facilitating skill transfer to clinical practice effectively at the lowest cost possible.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of a low-cost, locally designed simulation model (RAN) for flexible bronchoscope-guided tracheal intubation (FBTI) training, compared to a commercial airway part-task trainer. It aims to assess residents' skill acquisition, retention, and proficiency, promoting affordable simulation-based training.

The study follows a three-phase design:

Delphi Phase: Experts develop a standardized Global Rating Scale (GRS) for assessing FBTI skills through consensus.

Intermediate Phase: Piloting the tool with advanced trainees to ensure reliability and validity.

Main RCT Phase: PGY 1 and 2 residents, with no prior FBTI experience, are recruited from eight medical centers in Lebanon. Participants are randomly assigned to either the experimental (RAN model) or control (commercial trainer) group. Their FBTI skills are evaluated after training, and again at 3- and 6-month follow-ups, using the GRS on a high-fidelity airway simulator.

Data collection focuses on skill performance, with statistical models analyzing changes over time and between groups. The study aims to improve training accessibility while maintaining educational effectiveness.

ELIGIBILITY:
Phase 1: Expert committee Intermediate phase: Postgraduate fellows and residents from pulmonology and ENT, along with senior anesthesia residents Phase 2: Inclusion criteria include PGY 1 and 2 levels with no previous experience with FBTI and belonging to one of the eight prespecified medical centers. Any resident with prior exposure and experience with FBTI will be excluded.

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
A standardized global rating scale for FBTI skills assessment | Through the completion of the study phase 1; Immediately after the Delphi rounds are completed.
  The standardized global rating scale for FBTI skills assessment will be an adapted version of an existing global rating scale. It will be refined through Delphi rounds to achieve consensus in the first phase of this study.
Knowledge assessment | Baseline just before the Intervention; Directly after intervention; Three months after the intervention; and Six months after the intervention.
  Total score on the global rating scale (which will be the final output of the study phase 1: Delphi to improve and revise an available global rating scale). The higher the score on each item assessed the better the knowledge retained/acquired by the resident.
Technical skills assessment | Directly after intervention; Three months after the intervention; and Six months after the intervention.
  The technical skills will be assessed using the high-fidelity CASS simulator

CONTACTS AND LOCATIONS:
Overall Officials: Rony Al-Nawwar, MS, Study Director — Lebanese American University Medical Center - Rizk Hospital; Hanane Barakat, MD, Principal Investigator — Lebanese American University Medical Center - Rizk Hospital

IPD SHARING:
Plan to Share IPD: No